CLINICAL TRIAL: NCT02592291
Title: Mobile Health Self-Management and Support System for Chronic and Complex Health Conditions (Component 3)
Brief Title: Mobile Health Self-Management and Support System for Chronic and Complex Health Conditions
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Pittsburgh (Other)
Collaborators: Department of Health and Human Services (U.S. Federal Agency)
Responsible Party: Principal Investigator, Andi Saptono, Assistant Professor, University of Pittsburgh
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: STUDY19040337
Record Dates: First submitted 2015-10-23; First posted 2015-10-30 (Estimated); Last update posted 2025-10-03 (Actual); Status verified 2025-10

CONDITIONS: Spinal Cord Injuries; Cerebral Palsy; Spinal Dysraphism; Brain Injuries; Spina Bifida; Traumatic Brain Injury
Keywords: Mobile health; Apps; Applications; Smart phone; mHealth; Chronic and Complex Conditions; Self-Management; Self-Care
MeSH Terms: conditions — Spinal Cord Injuries; Cerebral Palsy; Spinal Dysraphism; Brain Injuries; Brain Injuries, Traumatic; Bronchiolitis Obliterans Syndrome

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- MHealth Group (Experimental): Participants randomized into this group will use the mHealth system throughout the study in conjunction with their standard of care
  Interventions: Device: MHealth
- Control (No Intervention): Participants randomized into this group will not use the mHealth system throughout the study, but will continue with their standard of care.

INTERVENTIONS:
Device: MHealth — The Mhealth system consists of a suite of apps to support participants manage their self-care and the clinician portal. Participants will use the system for 1 year.
  Arms: MHealth Group

SUMMARY:
This study will assess the benefits of using mobile health system designed for individuals with chronic and complex health conditions (such as those with Spinal Cord Injury,Cerebral Palsy, Spina Bifida, and Traumatic Brain Injury) to improve their wellness and self-management skills compared to those who receive standard of care only.

DETAILED DESCRIPTION:
Individuals with chronic and complex conditions such as those with spinal cord injury (SCI),Cerebral Palsy (CP), Spina Bifida (SB), and Traumatic Brain Injury (TBI), often require complex self-management routines to manage various needs such as bowel and bladder, skin integrity, and general health and wellness. Tasks such as self-catheterization, bowel regimens, skin checks, and routine administration of medications require consistent follow-through to prevent complications. Early detection and treatment of problems such as urinary tract infections (UTIs) or wounds, can prevent serious complications like osteomyelitis and sepsis which can result in hospitalization, death, and expensive medical care. The investigators have developed an innovative mobile health (mHealth) system aimed at improving self-management skills and preventing and detecting early signs of secondary medical complications. The system consist of a mobile health applications (apps), a clinician portal and a two-way secure communication system between the two. People with complex care regimens can use the apps to get reminders or cues to carry out their self care routines such as bowel/bladder routines, take medications, report success with their activities or new problems (e.g. new wound, UTI symptoms etc.), and track symptoms of depression. A clinician can use the portal to view the report and communicate with the users through a secure communication system that is embedded in the apps.

This study will assess the benefits of using the system in improving users' wellness and self-management skills compared to those who receive standard of care only.

ELIGIBILITY:
Inclusion Criteria:

1. 12 years or older.
2. have a diagnosis of a chronic and complex condition such as Spina Bifida, Spinal Cord Injury, Cerebral Palsy and Traumatic Brain Injury, etc.
3. live in a community setting (not within a residential facility that provides care to them).
4. pass all the functional screening tests which include basic usage of a smart phone, and impairment severity assessments

Exclusion Criteria:

1. Diagnosis of severe intellectual disability or severe and persistent psychiatric illness.
2. Failing all the screening tests due to severe impairments that cannot be accommodated by the mHealth system (for patient participants)

Min Age: 12 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 160 (Estimated)
Dates: Start 2019-10-01 (Actual); Primary Completion 2026-09 (Estimated); Study Completion 2026-09 (Estimated)

PRIMARY OUTCOMES:
Psychosocial Outcomes-Change of Self Management Skills Over Time as assessed by Self Management Questionnaire | At baseline and repeated on a schedule (approximately every three months) for up to 12 months
  Self management skill ratings measured at baseline, and approximately every three months for up to 12 months.
Psychosocial Outcomes-Change of Perceived Function and Satisfaction Over Time as assessed by Perceived Function and Satisfaction questionnaire. | At baseline and repeated on a schedule (approximately every three months) for up to 12 months
  Self ratings on perceived function and satisfaction questionnaire, assessed at baseline, and approximately every three months for up to 12 months.
Psychosocial Outcomes-Change of Quality of Life Over Time as assessed by Quality of Life questionnaire. | At baseline and repeated on a schedule (approximately every three months) for up to 12 months
  Quality of life ratings measured at baseline, and approximately every three months for up to 12 months.
Psychosocial Outcomes-Change of Function Ratings Over Time as assessed by Function or Physical Independence questionnaire. | At baseline and repeated on a schedule (approximately every three months) for up to 12 months
  Scale of Function measured at baseline, and approximately every three months for up to 12 months.
Psychosocial Outcomes- Change of Depressive Symptoms Over time as assessed by Depressive Symptoms questionnaire. | At baseline and repeated on a schedule (approximately every three months) for up to 12 months
  Questionnaire of Depressive symptoms administered at baseline, and approximately every three months for up to 12 months.
Medical Outcomes-Improvements in Preventable Conditions based on Medical Record Review | Through study completion, an average of 1 year.
  Medical record review of number of wounds, number of urinary tract infections and occurrences of sepsis.
Medical Outcomes-Improvements in Frequency of Health Care Utilization based on Medical Record Review and Questionnaire. | Through study completion, an average of 1 year.
  Medical Record Review and questionnaire on Number of hospitalizations, number of visits to emergency room and urgent care centers.
Medical Outcomes-Improvements in Length of Health Care Utilization based on Medical Record Review | Through study completion, an average of 1 year.
  Medical Record Review on Length of stay of hospitalizations.

SECONDARY OUTCOMES:
Change of Participants' experience using the mHealth system over time as assessed by questionnaire | At baseline and repeated on a schedule (approximately every three months) for up to 12 months)
  Questionnaire to assess participants subjective feelings about the use of the apps. This is for the MHealth group only.
Usage of the system as assessed by questionnaire and record review of the system usage (a built-in function in the system) | Through study completion, an average of 1 year.
  Questionnaire and review of usage record (a built-in function in the system) to measure the extent to which participants in the MHealth group consistently use the system to carry out their own self-management routines.
Cost of care | Through study completion, an average of 1 year.
  Estimated total cost of medical care.

CONTACTS AND LOCATIONS:
Overall Officials: Andi Saptono, Ph.D., Principal Investigator — University of Pittsburgh; Bambang Parmanto, Ph.D., Study Director — University of Pittsburgh; Brad E. Dicianno, M.D., Study Director — University of Pittsburgh
Locations (1):
- University of Pittsburgh, Pittsburgh, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Kryger MA, Crytzer TM, Fairman A, Quinby EJ, Karavolis M, Pramana G, Setiawan IMA, McKernan GP, Parmanto B, Dicianno BE. The Effect of the Interactive Mobile Health and Rehabilitation System on Health and Psychosocial Outcomes in Spinal Cord Injury: Randomized Controlled Trial. J Med Internet Res. 2019 Aug 28;21(8):e14305. doi: 10.2196/14305. PMID 31464189